CLINICAL TRIAL: NCT02909296
Title: Endoscopic Drainage of Collections After Pancreatic Surgery
Acronym: COLLECTOR
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: COLLECTOR
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic drainage

SUMMARY:
The pancreatic surgery causing some pancreatic collections. And in a number of case, this surgery can require a surgical resumption, a percutaneous drainage or an endoscopic drainage.

The endoscopic care of the treatment of pancreatic collections post-surgery is not yet standardized.

After failure of the medical treatment, the drainage of collections by echo-endoscopy was described.

There are not much series on this specific subject. Only 2 series contain more than 20 patients with 31 patients for the most important.

The timing and the technical choice of the endoscopic treatment as well as the long-term follow-up are not clear.

The purpose of this study is to estimate the success and the complications of the endoscopic drainage by echo-endoscopy according to the techniques of drainage and the timing of the endoscopic treatment.

The not estimated long-term follow-up will be also considered.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient having a pancreatic surgery complicated with a post-operative collection drained endoscopically

Exclusion Criteria:

* Contraindication surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having a pancreatic surgery complicated with a post-operative collection drained endoscopically
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Long-term evaluation of the risk of relapse | Up to 6 month
Timing of endoscopic drainage | Up to 3 month

SECONDARY OUTCOMES:
Immediate efficiency | Immediate post operative intervention

OTHER OUTCOMES:
Post surgery complications | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: CAILLOL Fabrice, MD, Principal Investigator — Institut Paoli-Calmettes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut PAOLI-CALMETTES — http://www.institutpaolicalmettes.fr